CLINICAL TRIAL: NCT00179491
Title: Study of the Therapeutic Effects of Intercessory Prayer (STEP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: John Templeton Foundation (Other); INTEGRIS Baptist Medical Center (Other); Medstar Health Research Institute (Other); Baptist Memorial Health Care Corporation (Other); Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2001-P-002125
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Artery Bypass Grafting Surgery
Keywords: coronary artery bypass grafting surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group 1 (Active Comparator): 604 patients received intercessory prayer after being informed they may or may not receive prayers (Group 1)
  Interventions: Behavioral: Intercessory Prayer
- 2 (No Intervention): 597 patients did not receive prayer after being informed they may or may not receive prayer (Group 2)
- Group 3 (Experimental): 601 patients received intercessory prayer after being informed they would receive it (Group 3).
  Interventions: Behavioral: Intercessory Prayer

INTERVENTIONS:
Behavioral: Intercessory Prayer — 14 days of intercessory prayer from 3 sites
  Arms: Group 1; Group 3

SUMMARY:
Intercessory prayer is widely believed to influence recovery from illness, but claims of benefits are not supported by well-controlled clinical trials. Prior studies have not addressed whether prayer itself or knowledge/certainty that prayer is being provided may influence outcome. We evaluated whether (1) receiving intercessory prayer or (2) being certain of receiving intercessory prayer was associated with uncomplicated recovery after coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
Intercessory prayer is widely believed to influence recovery from illness, but claims of benefits are not supported by well-controlled clinical trials. Prior studies have not addressed whether prayer itself or knowledge/certainty that prayer is being provided may influence outcome. We evaluated whether (1) receiving intercessory prayer or (2) being certain of receiving intercessory prayer was associated with uncomplicated recovery after coronary artery bypass graft (CABG) surgery.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or older
* Able to read or understand English

Exclusion criteria:

* Scheduled for emergent CABG (next available operating room slot)
* CABG more than 14 days after enrollment
* Other planned surgery within 30 days of CABG
* Minimally invasive CABG (non full sternotomy incisions)
* CABG with planned valve replacement, stent, angioplasty or carotid endarterectomy
* Or had ongoing chest pain or unstable angina, as defined by their physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1802 (Actual)
Dates: Start 1998-04; Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Whether receiving intercessory prayer was associated with uncomplicated recovery after coronary artery bypass graft (CABG) surgery. | 30 days

SECONDARY OUTCOMES:
Whether being certain of receiving intercessory prayer was associated with uncomplicated recovery after coronary artery bypass graft (CABG) surgery. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Benson, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Mind/Body Medical Institute